CLINICAL TRIAL: NCT01383642
Title: Physiology of Vestibular Dysfunction and Clinical Implications
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00035747-70
Record Dates: First submitted 2011-06-23; First posted 2011-06-28 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Dysfunction of Vestibular System; Accidental Falls; Frailty
MeSH Terms: conditions — Frailty | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- individuals age >=70
  Interventions: Other: No intervention, observational study

INTERVENTIONS:
Other: No intervention, observational study

SUMMARY:
Vestibular dysfunction is a known contributor to imbalance and fall risk, and may be a precursor to the frailty phenotype seen in the elderly population. A recent study found that vestibular dysfunction is common in the US population, and that the prevalence of this impairment increases steeply with age. However, it is unknown whether the aging process has global effects on the vestibular end-organ or whether specific structures, e.g. the semicircular canals or the otoliths, are selectively impaired. Moreover, the clinical implications of specific deficits of the vestibular end-organ are unclear. As such, the aims of this proposed research are: 1) to evaluate whether the normative aging process is predominantly associated with dysfunction of the semicircular canals (as measured by caloric and angular vestibulo-ocular reflex testing) or of the otoliths (as measured by vestibular-evoked myogenic potential (VEMP) testing); 2) to determine if there are any characteristic clinical features associated with the subtypes of vestibular dysfunction; and 3) to assess whether dysfunction of the semicircular canals or of the otoliths is associated with a higher risk of frailty and falls. The investigators plan to pursue these aims through a cross-sectional and prospective cohort study of a group of individuals age 70 and above. Vestibular physiologic tests will be administered to all study participants, and test results will be correlated with baseline clinical symptoms and frailty status as well as prospective one-year fall risk. A greater understanding of vestibular physiologic deficits and clinical implications in older individuals can inform the development of rational vestibular rehabilitation strategies that may more effectively mitigate the frailty phenotype and reduce fall risk.

ELIGIBILITY:
Inclusion Criteria:

* Participant's age is 70 years and over?
* Participant is willing and able to give informed consent?

Exclusion Criteria:

* Participant has diabetes mellitus
* Participant has blindness, limited neck range of motion or cervical spine instability

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: community-dwelling adults age >70
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
vestibular function | baseline

SECONDARY OUTCOMES:
Number of participants who report one or more falls in a one-year follow-up period | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States